CLINICAL TRIAL: NCT01010620
Title: Screening Protocol for the Evaluation of Research Participants
Brief Title: Screening Protocol for Research Participants
Acronym: ScreenProt
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Deanna L. Kelly, PharmD., BCPP Professor of Psychiatry Director, Treatment Research Program (TRP), University of Maryland, Baltimore
Other Study IDs: HP-00043664; MPRC #412; NIDA #444
Record Dates: First submitted 2009-07-08; First posted 2009-11-10 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Substance Abuse; Cocaine Abuse; Tobacco Use Disorder
Keywords: screening; research participation; substance abuse; Schizophrenia; nicotine; Healthy; cigarettes; smoking; marijuana; cocaine
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders; Cocaine-Related Disorders; Tobacco Use Disorder; Smoking; Marijuana Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening: Screening Assessment battery. Specific to study(or studies) the individual is screening for.
  Interventions: Behavioral: Various Screening psychiatric and medical assessments

INTERVENTIONS:
Behavioral: Various Screening psychiatric and medical assessments — Possibly blood draws, urine samples, toxicology screens, computer-based and written psychological, psychiatric, and behavioral questionnaires and assessments.

SUMMARY:
The Screening Protocol is a system devised to evaluate potential research participants for National Institute on Drug Abuse/Maryland Psychiatric Research Center (NIDA/MPRC) studies.

DETAILED DESCRIPTION:
The MPRC/NIDA collaborative research program attempts to: elucidate the nature of serious mental illnesses, drug abuse and addiction; determine the potential use of new therapies, both pharmacological and psychosocial; and decipher the long-term effects of drugs of abuse on the development, maturation, function, and structure of the brain and other organ systems. In support of this work, the scientific goal of this screening protocol is to assess potential research participants' eligibility for research studies. Screening will include medical and psychological tests and procedures. The data collected during screening are a unique and valuable source of information that aids in the research mission. Therefore, a secondary goal of this protocol is to obtain data that characterizes the population of subjects contacting NIDA about research participation and to analyze data so obtained, such as that on the prevalence and consequences of HIV/AIDS, viral hepatitis, and related diseases and issues of selection and sample bias in clinical research.

The screening process will be done in two stages, a telephone interview and an in-person evaluation. The telephone interview will last approximately 20 minutes and be conducted solely via the NIDA call center. Answers provided during the phone interview will indicate whether a caller is eligible for in-person screening. Those who appear eligible will be given an appointment at either NIDA or MPRC. This protocol pertains only to the in-person participants at MPRC. Written informed consent will be obtained when the person arrives. The screening process can involve up to 5 visits to MPRC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to read and understand and answer questions posed.

Exclusion Criteria:

* Inability to provide valid informed consent
* Below Age 18, and above age 64.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Population will see an advertisement in the community and call the NIDA call center. If they appear to meet the qualifications for one or more NIDA/MPRC studies, they will be scheduled to be screened.
Sampling Method: Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment of participants into NIDA/MPRC protocols. | 5 years

SECONDARY OUTCOMES:
Demographic characterization of drug users, non-users, and individuals with serious mental illnesses contacting NIDA/MPRC about research participation | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D., BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States